CLINICAL TRIAL: NCT06604897
Title: Effectiveness of Entresto (Sacubitril/Valsartan) to Blood Pressure Control in Japanese Patients With Hypertension: the Database Analysis of Electronic Medical Records
Brief Title: Effectiveness of Entresto (Sacubitril/Valsartan) in Japanese Patients With Hypertension
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CLCZ696AJP04
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Sacubitril/Valsartan Cohort: Adult patients with essential hypertension who were prescribed sacubitril/valsartan.
- Conventional Drug-control Cohort: Adult patients with essential hypertension who were prescribed angiotensin-converting enzyme inhibitor/angiotensin receptor blocker (ACEi/ARB).

SUMMARY:
This study is a non-interventional, secondary use of data, retrospective, cohort study, and the data to be extracted in this study will be used as secondary use of collected patient information in the database (Japan Medical Data Survey [JAMDAS]) owned by M3 Inc. JAMDAS is a database that aggregates medical information and is constructed mainly from electronic medical record information of general practices, allowing real-time extraction of information entered in medical records, such as prescription status including drug switching and continuation, laboratory values, clinical evaluation scores, and comorbidities, etc.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed with essential hypertension (International Classification of Diseases [ICD]-10 code: I10) on the index date.
2. Patients for whom data for the 6 months prior to the index date can be extracted as baseline data.
3. Patients for whom blood pressure (BP) data can be extracted between weeks 8 and 12 after the index date.
4. Patients whose BP data can be extracted on the index date.
5. Patients whose BP value at baseline was 140/90 millimeters of mercury (mmHg) or higher.
6. Patients with the prescription of 100 milligrams (mg) or 200 mg once daily as 100 mg or 200 mg tablets on the index date.

Exclusion criteria:

1. Women with a record of pregnancy-related diagnoses, drugs, or medical procedures before or after the index date, or a record of delivery- or abortion-related diagnoses, drugs, or medical procedures after the index date.
2. Prescription of concomitant angiotensin-converting enzyme inhibitor (ACEi); Anatomical Therapeutic Chemical (ATC) code: C09A on, after, or in the 2 days before the index date.
3. Patients diagnosed with angioedema: ICD-10: D84.1 under prescription of ACEi or angiotensin receptor blocker (ARB); ATC code: C09C.
4. Patients diagnosed with diabetes and under treatment with aliskiren fumarate on the index date.
5. Patients with severe impaired liver functions with Child-Pugh classification C.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1405 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients Achieving the Guideline-recommended Blood Pressure (BP) | Up to approximately 12 weeks (the BP measurement timepoint closest to 8 weeks between weeks 8 and 12)
  The Japanese Society of Hypertension Guidelines for the Management of Hypertension (JSH 2019) will be used to establish systolic and diastolic blood pressure goals.

SECONDARY OUTCOMES:
Percentage of Patients Achieving the Guideline-recommended Blood Pressure (BP) per BP Category | Up to approximately 12 weeks (the BP measurement timepoint closest to 8 weeks between weeks 8 and 12)
  The Japanese Society of Hypertension Guidelines for the Management of Hypertension (JSH 2019) will be used to establish systolic and diastolic blood pressure goals.
  BP categories:
  * Grade I: 140-159/90-99 millimeters of mercury (mmHg)
  * Grade II: 160-179/100-109 mmHg
  * Grade III: 180/110 mmHg or greater
Percentage of Patients Achieving the Guideline-recommended BP Categorized by Number of Antihypertensive Medicines Taken Before Starting Sacubitril/Valsartan | Up to approximately 12 weeks (the BP measurement timepoint closest to 8 weeks between weeks 8 and 12)
  The Japanese Society of Hypertension Guidelines for the Management of Hypertension (JSH 2019) will be used to establish systolic and diastolic blood pressure goals.
  Number of antihypertensive medicines taken before starting sacubitril/valsartan categories: 0, 1, 2, 3-4, and 5 or more.
Percentage of Patients Achieving the Guideline-recommended BP Categorized by Antihypertensive Drug Classes Prescribed With Sacubitril/Valsartan | Up to approximately 12 weeks (the BP measurement timepoint closest to 8 weeks between weeks 8 and 12)
  The Japanese Society of Hypertension Guidelines for the Management of Hypertension (JSH 2019) will be used to establish systolic and diastolic blood pressure goals.
  Antihypertensive drug classes include:
  * Calcium channel blockers (CCB)
  * Angiotensin-converting enzyme (ACE) inhibitors
  * Angiotensin receptor blockers (ARBs)
  * Diuretics
  * Alpha and beta blockers
  * Alpha-beta blockers
  * Aldosterone blockers
  * Renin inhibitors
  * Compounding agents
Percentage of Patients Achieving the Guideline-recommended BP Categorized by Patient Characteristics | Up to approximately 12 weeks (the BP measurement timepoint closest to 8 weeks between weeks 8 and 12)
  The Japanese Society of Hypertension Guidelines for the Management of Hypertension (JSH 2019) will be used to establish systolic and diastolic blood pressure goals.
  Patient characteristics include, but are not limited to, age, gender, body mass index (BMI), comorbidities, and combinations of comorbidities.
Number of Patients Categorized by Place of Residence | Baseline
Height | Baseline
Weight | Baseline
Number of Patients Categorized by Comorbidities | Baseline
  Comorbidities include:
  * Heart disease
  * Diabetes
  * Dyslipidemia
  * Renal disease
  * Cerebrovascular disease
  * Other, specify
Relative Contribution of Baseline Characteristics in Achieving the Guideline-recommended BP | Up to approximately 12 weeks (the BP measurement timepoint closest to 8 weeks between weeks 8 and 12)
  The Japanese Society of Hypertension Guidelines for the Management of Hypertension (JSH 2019) will be used to establish systolic and diastolic blood pressure goals.
  Multivariate logistic regression analysis will be used to determine the association of the following variables in achieving the guideline-recommended BP.
  * Age
  * Gender
  * Comorbidities
  * Body mass index (BMI)
  * BP category at index date
  * Number of classes of antihypertensive medicines taken before starting sacubitril/valsartan
Persistence on Sacubitril/Valsartan | Up to 16 weeks
  Proportion of patients remaining on treatment with sacubitril/valsartan and proportion of patients permanently discontinuing sacubitril/valsartan during the study.
Number of Episodes of Hypotension-related Events | Up to 16 weeks
  Hypotension-related events include:
  * Orthostatic hypotension
  * Postural hypotension
  * Secondary orthostatic hypotension
  * Hypertension due to the drugs
  * Episodic hypotension
  * Hypotension
  * Vertigo
  * Feeling dizzy
  * Dizziness
  * Sudden dizziness
  * Syncope
Number of Episodes of Renal Events | Up to 16 weeks
  Renal events include:
  * Renal diseases
  * Chronic kidney disease (CKD)
  * Estimated glomerular filtration rate (eGFR) reduction of 40% or more
Number of Episodes of Dehydration-related Events | Up to 16 weeks
  Dehydration-related events include:
  * Dehydration
  * Isotonic dehydration
Number of Episodes of Diuresis-related Events | Up to 16 weeks
  Diuresis-related events include:
  * Polyuria
  * Idiopathic polyuria
  * Frequent urination
  * Nocturnal polyuria
  * Nocturia
Number of Episodes of Edema or Angioedema-related Events | Up to 16 weeks
  Edema or angioedema-related events include:
  * Angioneurotic edema
  * Quincke's edema
Percentage of Patients Treated With Sacubitril/Valsartan Achieving the Guideline-recommended BP Compared to the Percentage of Patients Treated With Angiotensin-converting Enzyme Inhibitor/Angiotensin Receptor Blocker (ACEi/ARB) | Up to approximately 12 weeks (the BP measurement timepoint closest to 8 weeks between weeks 8 and 12)
  The Japanese Society of Hypertension Guidelines for the Management of Hypertension (JSH 2019) will be used to establish systolic and diastolic blood pressure goals.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States